CLINICAL TRIAL: NCT05901259
Title: The Exopulse Mollii Suit Study - a Database for Routine Follow-up of Clinical Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Exoneural Network AB (Industry)
Responsible Party: Sponsor
Other Study IDs: CIV-22-08-040366
Record Dates: First submitted 2023-05-29; First posted 2023-06-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Palsy; Multiple Sclerosis; Stroke; Spinal Cord Injuries; Neurologic Disorder
MeSH Terms: conditions — Cerebral Palsy; Multiple Sclerosis; Stroke; Spinal Cord Injuries; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Exopulse Mollii Suit — The registry is designed to demonstrate the impact of Exopulse Mollii Suit on improvement of muscle relaxation, muscle activation, local blood circulation and/or chronic pain relief. The subjects included use the suit for 60 minutes every other day, unless other is specified by the Investigator, in their home environment for up to a maximum of 12 consecutive weeks. Qualitative and quantitative measures will be collected at baseline (T0), after 60 minutes stimulation (T1), after 4 weeks (T4) and at the end of the 12-week intervention period (T12).

SUMMARY:
The objective is to explore the potential short and long-term impact of the Exopulse Mollii Suit on subjects with CP, MS, stroke, SCI or other neurological disorders which may cause such types of symptoms, and to identify high responders among the sub-categories of the diagnoses. The primary endpoint will be improvement on the Berg/Pediatric Balance Scale (BBS) as a measurement of balance and risk of falls.

DETAILED DESCRIPTION:
The registry is designed to demonstrate the impact of Exopulse Mollii Suit on improvement and relaxation of muscles, muscle activation, local blood circulation and chronic pain relief.

The subjects will serve as their own control and the data will be collected before, during and after the treatment period. As the electrical stimulation from the suit usually is above the level of sensation, the study participant cannot be blinded to the treatment.

To prevent bias, multiple investigators will be collecting the data and only standardized and validated methods will be used. All investigators will be trained on the measurements prior to the registry start.

Additionally, all investigators are trained and certified in the Exopulse method, and the generic stimulation settings are selected according to a standardized matrix based on the subjects' age and level of impairment.

Re-assessments during scheduled visits are part of normal routine and use. The decision whether the subjects will be enrolled in the registry is separated from the subject's decision to use the device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CP, MS, stroke, spinal cord injury or other neurologic disorder that may cause such type of symptoms.
* Diagnosed >6 months prior to inclusion in case of MS, stroke, or SCI
* Give written informed consent
* Cognitively able to understand and follow verbal and/or written instructions
* A minimum age of 2 years

Exclusion Criteria:

* Any of the contraindications listed in the instructions for use of the Exopulse Mollii Suit
* Being introduced to any new medication affecting the neuromuscular activity during the study period
* Using botulinum toxin <3 month before or during the study period
* Subjects <100 cm and <13 kg
* Subjects >205 cm and >115 kg

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects over 2 years of age diagnosed with CP, MS, stroke, spinal cord injury or other neurologic disorder that may cause such type of symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Berg's Balance Scale | To be assessed at baseline, after 60 minutes stimulation (T1), after 4 weeks (T4) and at the end of the 12-week intervention period (T12).
  Change in balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in Patients with Multiple Sclerosis (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.

SECONDARY OUTCOMES:
Timed Up and Go (TUG), if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  Change in walking velocity will be assessed with TUG. Patients have to stand up from a chair when they hear the verbal instruction "go", walk a distance of 3 meters, turn around, walk back to the chair and sit down. Timing starts with the verbal instruction "go' and stops when the patients return to the seated position. The score consists of the time taken to complete the test activity, measured in seconds.
10 m Walk Test, if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  The 10mWT is used to assess the change in walking speed in meters/second (m/s) over a short distance.
Wolf Motor Function Test, if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  The change in upper motor ability will be assess with WMFT. WMFT is a quantitative measure of upper extremity motor ability through timed and functional tasks.
Numeric Rating Scale (NRS), if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  The change in pain will be assess with NRS. NRS measures the subjective intensity of pain, where 0=no pain and 10=worst possible pain.
EQ-5D-5L, if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  The change in quality of life will be assessed with EQ-5D, which is an instrument which evaluates the generic quality of life. Designed as a self-completion questionnaire, it embodies two components, a health state description followed by an evaluation.The respondent classifies his or her prevailing state of health by selecting one of three different levels of problem severity within each of five health domains.
Fibromyalgia Impact Questionnaire (FIQ), if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  The change in function will be assessed with FIQ. The FIQ evaluates the function, overall impact and symptoms of fibromyalgia over the last 7 days.
  The FIQ is composed of 10 items. The first item contains 11 questions related to physical functioning - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression.
Quebec Back Pain Disability Scale, if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  The change in back pain will be assessed with Quebec Back Pain Disability Scale. The Quebec back pain disability scale (QBPDS) is a condition-specific questionnaire which measures the level of functional disability for patients with low back pain. The scoring is done by counting every digit, circled by the patient. The end score will be between 0 (no limitation) and 100 (totally limited).
Near Infrared Spectroscopy (NIRS), if applicable for the patient | To be assessed at baseline, immediately after 60 minutes stimulation (T1), 4 weeks after first visit (T4) and at the end of the 12-week intervention period (T12).
  The change in tissue oxygenation index will be evaluated using NIRS technology. A wireless device PortaMon (Artinis Medical Systems, The Netherlands)- is designed for this purpose, it consists of three light emitting diodes, each sending two wavelengths and four channels to measure tissue oxygenation index.

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Westerlund, Phd, Principal Investigator — Exoneural Network AB
Locations (1):
- Exoneural Network Ab, Bergshamra, Stockholm County, Sweden